CLINICAL TRIAL: NCT03690973
Title: Evaluation of Bone Changes of The Extraction Sockets After Immediate Implant or Socket Preservation With or Without Surgical Flap in The Aesthetic Zone "Randomized Controlled Clinical Trial"
Brief Title: Evaluation of Bone Changes After Immediate Implant Placement or Socket Preservation With or Without Surgical Flap in The Aesthetic Zone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Shaarawi, Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: perio2018
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Alveolar Socket Preservation
Keywords: Bone graft; Immediate dental implant; Flap; Flapless
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Masking Description: single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Alveolar socket preservation with graft and flap surgery (Active Comparator)
  Interventions: Drug: Alveolar socket preservation with graft and flap surgery
- Immediate implant placement with bone using flapless surgery (Experimental)
  Interventions: Device: Immediate implant placement with bone using flapless surgery
- Immediate implant placement with bone and flap surgery (Experimental)
  Interventions: Device: Immediate implant placement with bone using flap surgery
- Alveolar socket preservation with graft and flapless surgery (Experimental)
  Interventions: Drug: Alveolar socket preservation with graft and flapless surgery

INTERVENTIONS:
Drug: Alveolar socket preservation with graft and flap surgery — Alveolar socket preservation with xenogenic bone graft and flap surgery
  Arms: Alveolar socket preservation with graft and flap surgery
Device: Immediate implant placement with bone using flapless surgery — Immediate implant placement with xenogenic bone graft using flapless surgery
  Arms: Immediate implant placement with bone using flapless surgery
Device: Immediate implant placement with bone using flap surgery — Immediate implant placement with xenogenic bone graft using flap surgery
  Arms: Immediate implant placement with bone and flap surgery
Drug: Alveolar socket preservation with graft and flapless surgery — Alveolar socket preservation with xenogenic bone graft and flapless surgery
  Arms: Alveolar socket preservation with graft and flapless surgery

SUMMARY:
The amount of hard tissue resorption following tooth extraction involves prosthetically driven implant placement; therefore, the development of ridge preservation techniques that result in less alveolar bone loss is of great interest, Alveolar ridge preservation are indicated to decrease the loss of ridge volume that follows tooth extraction.However, they do not prevent bone resorption because, depending on the technique.The protocol of placing implants immediately upon tooth extraction has been introduced into clinical practice which aims to preserve the socket from resorption, also immediate implant satisfy the patient as it decrease the time for crown insertion in addition to that it has a good survival.There is not adequate research data to clearly demonstrate that flapless socket preservation techniques are superior to techniques that involve raising a flap, but an animal study reported that the detachment of the periosteum from the buccal site of the ridge leads to an increase of the resorption rate, resulting in an increase of the ridge resorption

DETAILED DESCRIPTION:
Socket preservation procedures have been performed to preserve hard and soft tissue volume, which can be partially lost after tooth removal. These procedures allow for wider and longer implant placement compared with non-augmented sockets and reduce the need for simultaneous augmentation procedures at the time of implant placement.It is expected that immediate implant avoid crestal resorption in the fresh extraction socket in humans also immediate installation at the time of extraction offers potential advantages for both practitioners and patients. It allows a decrease in treatment time and may result in an increase in patient satisfaction.Also it is expected that flapless procedure include maintenance of the buccal keratinized gingival , and prevention of alterations to the gingival contours and migration of the mucogingival junction that are often experienced after raising a flap

ELIGIBILITY:
Inclusion Criteria:

1. Age: Above 18 years.
2. Patients with single non-restorable teeth in anterior or premolar area.
3. Patients with adequate bone volume for the dental implant procedure.
4. Patients with good oral hygiene
5. Patient consent approval and signing.

Exclusion Criteria:

1. Heavy smokers.
2. Systemic disease that contraindicates surgical implant placement
3. Presence of any acute pathosis at the site of surgery.
4. Patients with thin alveolar ridge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Bone volume changes | 1 year
  volumetric bone changes by cone-beam computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Amr Zahran, Phd, Study Chair — Cairo University; Ahmed Reda, Phd, Study Chair — Cairo University
Locations (1):
- Amr Mohamed Shaarawi, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
I will check with my study chair

REFERENCES:
- [Background] Aimetti M, Manavella V, Corano L, Ercoli E, Bignardi C, Romano F. Three-dimensional analysis of bone remodeling following ridge augmentation of compromised extraction sockets in periodontitis patients: A randomized controlled study. Clin Oral Implants Res. 2018 Feb;29(2):202-214. doi: 10.1111/clr.13099. Epub 2017 Nov 17. PMID 29148597
- [Background] Tonetti MS, Cortellini P, Graziani F, Cairo F, Lang NP, Abundo R, Conforti GP, Marquardt S, Rasperini G, Silvestri M, Wallkamm B, Wetzel A. Immediate versus delayed implant placement after anterior single tooth extraction: the timing randomized controlled clinical trial. J Clin Periodontol. 2017 Feb;44(2):215-224. doi: 10.1111/jcpe.12666. Epub 2017 Jan 31. PMID 27978602